CLINICAL TRIAL: NCT00178646
Title: Comparative Efficacy of Three Preparations of Botox-A in Treating Spasticity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Gerard Francisco, Clinical Professor and Chairman - Physical Medicine and Rehabilitation, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-01-103
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Stroke; Brain Injuries; Spasticity
Keywords: Stroke; Brain Injuries; Spasticity; Botulinum Toxins
MeSH Terms: conditions — Stroke; Brain Injuries; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 - Low Volume, High Dose (Experimental): Botox (onabotulinumtoxinA), 150 units prepared as 100 units per 1 ml of preservative-free normal saline
  Interventions: Drug: Botox
- 2 - High Volume, High Dose (Active Comparator): Botox (onabotulinumtoxinA), 150 units prepared as 50 units per 1 ml of preservative-free normal saline
  Interventions: Drug: Botox
- 3 - High Volume, Low Dose (Other): Botox (onabotulinumtoxinA), 75 units prepared as 25 units per 1 ml of preservative-free normal saline
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — Botox 75-150 units, single treatment only
  Other Names: generic name: botulinum toxin type A

SUMMARY:
The study seeks to compare the effectiveness of three preparations of BOTOX-A® in treating muscle tightness and spasms in the feet and ankles of people with stroke.

DETAILED DESCRIPTION:
Spasticity is one of the most debilitating complications of neurologic conditions, such as stroke, brain injury, spinal cord injury, cerebral palsy, and multiple sclerosis. Although the exact pathophysiology is unknown, it is believed to result from an imbalance of ascending excitatory influences on and descending inhibitory components of the central nervous system. Clinically, spasticity manifests as abnormally increased muscle tone, associated with loss of range of motion, increased muscle stretch reflexes, clonus, weakness, and incoordination. If inadequately treated, spasticity leads to more disability and increase health care costs. Common complications of inadequately treated spasticity include joint and muscle contracture, pain, difficulty with performing activities of daily living and hygiene, and impaired transfers and ambulation.

Acquired brain injuries (ABI), including stroke, traumatic brain injury, and encephalopathy, often lead to long-term impairments, including spasticity. In severe cases, spasticity is difficult and frustrating to treat in this patient population, since the individuals may not tolerate the side effects of conventional therapies because of ABI-related deficits in arousal and cognition. Systemic medications, such as baclofen and tizanidine, are effective in controlling spasticity; however, they may also cause sleepiness and drowsiness, and impair memory and thinking processes---adverse effects that individuals with ABI may not tolerate.

Thus, "local" treatments, such as neurolysis and chemodenervation using botulinum toxin, have become superior treatment options in individuals with ABI, since they are devoid of the usual side effects of systemic medications. They are also effective in controlling spasticity, yet they do not impair arousal and cognition. The medical literature is replete with reports of the efficacy of botulinum toxin-A in the management of spasticity. Thus, the current challenge for clinicians and researchers at this time is to find ways to further enhance the efficacy of botulinum toxin. One way to achieve this is by exploiting certain properties of the toxin. Animal studies and clinical experience have shown that the effects of the drug is dose-dependent. One other property is the flexibility in preparing the volume of drug injected. Since botulinum toxin, as it is currently available (as BOTOX-A®) in the United States, requires reconstitution with preservative-free saline, there is flexibility for clinicians to manipulate the volume of solution that will be administered, without altering the dose.

We recently completed a trial comparing the effects of two volume preparations of BOTOX-A® on wrist and finger flexor spasticity of individuals with ABI. One group of patients received BOTOX-A® prepared as 100 units/cc, while another received BOTOX-A® prepared as 50 units/cc. Although there was no statistically significant difference between the two groups, there was a trend in favor of the group that received the higher volume, i.e.; they appeared to improve more based on decrease in muscle tone (measured by the Modified Ashworth Scale). This was compared by the clinician's global impression that the high volume group improved more. The latter measure achieved statistical significance. One possible reason for the absence of statistical significance was that the "high" volume (50 units/cc) was not high enough. Thus, we are proposing this study to investigate the comparative effects of three preparations of BOTOX-A®.

ELIGIBILITY:
Inclusion Criteria -

* Spasticity resulting from ABI (stroke, including vascular malformations, traumatic brain injury)
* Ashworth Score (resting) of at least 2 of the primary ankle plantarflexor (gastrocnemius)
* Onset of primary illness at least six months prior to study inclusion
* At least 12 years of age

Exclusion Criteria -

* Hypersensitivity or allergy to botulinum toxin
* History of myasthenia gravis or other neuromuscular disease
* Current use of aminoglycosides
* Botulinum toxin or phenol injection to study limb within six months prior to recruitment
* Current use of other spasmolytic drug, such as diazepam, baclofen, dantrolene, tizanidine
* Presence of contracture or significant muscle atrophy
* Pregnancy

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2002-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerard E Francisco, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Kessler Institute for Rehabiliation, West Orange, New Jersey
  - Memorial Hermann Hospital, Houston, Texas

REFERENCES:
- [Background] Francisco GE, Boake C, Vaughn A. Botulinum toxin in upper limb spasticity after acquired brain injury: a randomized trial comparing dilution techniques. Am J Phys Med Rehabil. 2002 May;81(5):355-63. doi: 10.1097/00002060-200205000-00007. PMID 11964576

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 were enrolled but 32 started, and this is because one participant who enrolled decided not to start the study.
Groups:
- Low Volume, High Dose: Botox, 150 units prepared as 100 units/ml
  Botox: Botox 75-150 units, single treatment only
- High Volume, High Dose: Botox 150 units, prepared as 50 units/ml.
  Botox: Botox 75-150 units, single treatment only
- High Volume, Low Dose: Botox 75 units, prepared as 25 units/ml.
  Botox: Botox 75-150 units, single treatment only
Period: Overall Study
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Started | 12 | 9 | 11
Completed | 12 | 8 | 10
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Low Volume, Low Dose: Botox 75 units, prepared as 25 units/ml.
  Botox: Botox 75-150 units, single treatment only
- Total: Total of all reporting groups
Arm/Group | Low Volume, High Dose | High Volume, High Dose | Low Volume, Low Dose | Total
Number analyzed (Participants) | 12 | 9 | 11 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 9 | 11 | 32
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 10 | 5 | 8 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Spastic Hypertonia as Measured by the Ashworth Scale
Description: The Ashworth Scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Score on the Ashworth scores ranges from 0-4, with 4 being the worst:
  0 - No increase in muscle tone
  1. - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  2. - More marked increase in muscle tone through most of the range of motion, but affected limb easily flexed
  3. - Considerable increase in muscle tone, passive movement difficult
  4. - Limb in flexion or extension
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 12 | 9 | 11
score on a scale | 2.4 [2 to 3] | 2.33 [2 to 3] | 2.36 [1 to 3]

2. Primary Outcome: Spastic Hypertonia as Measured by the Ashworth Scale
Description: The Ashworth Scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. Score on the Ashworth scores ranges from 0-4, with 4 being the worst:
  0: No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  2. More marked increase in muscle tone through most of the range of motion, but affected limb easily flexed
  3. Considerable increase in muscle tone, passive movement difficult
  4. Limb in flexion or extension
Time Frame: Four weeks
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Low Volume, High Dose: Low volume, High Dose:
  Botox, 150 units prepared as 100 units/ml
  Botox: Botox 75-150 units, single treatment only
- High Volume, High Dose: High volume, High Dose:
  Botox 150 units, prepared as 50 units/ml.
  Botox: Botox 75-150 units, single treatment only
- High Volume, Low Dose: HIgh Volume, Low Dose:
  Botox 75 units, prepared as 25 units/ml.
  Botox: Botox 75-150 units, single treatment only
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 12 | 9 | 11
score on a scale | 2.42 [2 to 3] | 2.56 [2 to 3] | 2.36 [1 to 3]

3. Primary Outcome: Spastic Hypertonia as Measured by the Ashworth Scale
Description: as for outcome 2
Time Frame: Eight Weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 12 | 9 | 11
score on a scale | 1.42 [0 to 3] | 0.77 [0 to 2] | 1 [0 to 2]

4. Primary Outcome: Spastic Hypertonia as Measured by the Ashworth Scale
Description: as for outcome 2
Time Frame: Twelve Weeks
Population: Data for this outcome measure were not collected for 2 in the Low volume High Dose arm, 1 in the High volume High Dose arm, and 1 in the High Volume Low Dose arm.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 10 | 8 | 10
score on a scale | 1.3 [0 to 2] | 1 [0 to 2] | 1.7 [1 to 3]

5. Primary Outcome: Spastic Hypertonia as Measured by the Ashworth Scale
Description: as for outcome 2
Time Frame: Sixteen Weeks
Population: Data for this outcome measure were not collected for 1 in the High volume High Dose arm and 1 in the High Volume Low Dose arm.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 12 | 8 | 10
score on a scale | 1.42 [0 to 2] | 1.13 [1 to 2] | 1.1 [0 to 2]

6. Secondary Outcome: Range of Motion as Measured by Goniometry
Description: This outcome reports the angle formed during ankle dorsiflexion by an imaginary line drawn on the outer side of the leg with an imaginary line drawn on the outside of the foot. The angle changes as the ankle is curled up (dorsiflexed) or down (plantarflexed). Many people with stroke develop muscle tightness (a condition called spasticity) or contracture, which leads to ankle plantarflexion and results in a "foot drop" appearance and limits range of motion.
  When the ankle is neutral and the foot is flat, the angle between the leg and the foot is roughly a right angle, and this neutral position is indicated as 0 degrees from the neutral position. If the foot is below the neutral position during maximum ankle dorsiflexion, then the angle reported is the number of degrees below the neutral position (reported as a negative value). If the foot is above the neutral position, then the angle reported is the number of degrees above the neutral position (positive value).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 12 | 9 | 11
degrees | -9.42 (5.42) | -6.56 (9.96) | -19.64 (13.90)

7. Secondary Outcome: Range of Motion as Measured by Goniometry
Description: as for outcome 6
Time Frame: 8 weeks
Population: Data were not collected for on in the Low volume, High Dose arm, one in the High volume, High Dose arm, and one in the High Volume, Low Dose arm.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Low Volume, High Dose | High Volume, High Dose | High Volume, Low Dose
Number analyzed (Participants) | 11 | 8 | 10
degrees | -1.82 (6.82) | 2.25 (8.08) | -2.30 (6.57)

ADVERSE EVENTS:
Time Frame: Four months
Arm/Group | Low Volume, High Dose | High Volume, High Dose | Low Volume, Low Dose
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 2/9 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Volume, High Dose (N=12) | High Volume, High Dose (N=9) | Low Volume, Low Dose (N=11)
Visual Change (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Altered Mental Status (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bowel urgency (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased Salivation (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes